CLINICAL TRIAL: NCT00606346
Title: A Multicenter, Prospective, Long-term, Observational Registry of Pediatric Patients With Inflammatory Bowel Disease
Acronym: DEVELOP
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013912; C0168Z02 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; Inflammatory Bowel Diseases
Keywords: Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; Inflammatory Bowel Diseases; Immunomodulators; infliximab; TNF-alpha
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti TNF therapy including infliximab: Treatments will be prescribed according to investigator judgement.
  Interventions: Biological: Anti TNF therapy including infliximab
- No Biologics: Treatments will be prescribed according to investigator judgement.
  Interventions: Drug: No Biologics

INTERVENTIONS:
Biological: Anti TNF therapy including infliximab — Treatments will be prescribed according to investigator judgement.
  Groups: Anti TNF therapy including infliximab
Drug: No Biologics — Treatments will be prescribed according to investigator judgement.
  Groups: No Biologics

SUMMARY:
The purpose of this study is to evaluate the long-term safety and clinical status of pediatric patients with Inflammatory Bowel Disease (IBD). Particular attention will be directed to recording safety outcomes reported in association with infliximab and other prescribed IBD therapies. In addition, information on disease status and quality of life will be collected.

DETAILED DESCRIPTION:
This registry study will include volunteer pediatric patients: approximately 2,000 pediatric patients with Crohn's Disease who have been treated with infliximab and approximately 2,000 pediatric patients with Crohn's Disease who have received therapies other than infliximab. Approximately 1,000 pediatric patients with Ulcerative Colitis or Indeterminant Colitis will also be enrolled. All patient treatments for IBD will be decided by the treating physicians in consultation with their patients based on usual clinical practice. Patient information will be collected at the time of enrollment and every 6 months for approximately 20 years. Data collection will include disease characteristics, IBD medications, safety assessments to include adverse events. Patients will also be asked to complete a brief questionnaire describing school and/or work attendance in order to assess quality of life. Some patients may be asked to participate in a substudy that will evaluate blood levels of formation of proteins that may develop after treatment with infliximab. A small amount of additional blood may be taken at the time of a routine blood draw that is part of a patient's routine medical care as determined by a treating physician. There are three studies as part of the post marketing requirement for IBD - C0168Z02, REMICADEPIB4002 and REMICADEPIB4003. There is one combined database for these protocols and analyses are performed using the aggregate data. All reports and publications will be generated from the combined database. No study agents will be administered in this registry. All patients will receive standard-of-care treatments prescribed by the patient's physician.

ELIGIBILITY:
Inclusion Criteria:

C0168Z02 - Confirmed diagnosis of Crohn's disease, Ulcerative Colitis, or Indeterminate Colitis for at least 2 months The parent/legal guardian must be capable of providing written informed consent, and assent should be obtained from the child according to local regulations (age at which assent is given may vary by the IRB or EC).

The patient's physician expects the patient to be scheduled for a medical encounter (and/or other direct contact) at least every 6 months, as part of their usual care, at the time of enrollment.

REMICADEPIB4002 and REMICADEPIB4003: Confirmed diagnosis of Crohn's disease or Ulcerative Colitis for at least 2 months

Exclusion Criteria:

C0168Z02: 17 years of age or older, with the exception of patients who participated in the Sponsor's conducted pediatric IBD clinical trials.

Have other Crohn's-like diseases that are associated with genetic diseases (eg, glycogen storage disease).

The patient and parent/guardian are not able to adhere to the protocol requirements.

Are participating in any clinical trial for an investigational agent that is not commercially available.

REMICADEPIB4002 and REMICADEPIB4003: Less than 6 years of age or 17 years of age or older.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a registry of pediatric patients with IBD (e.g., CD, UC, or IC in C0168Z02 and CD in REMICADEPIB4002 and REMICADEPIB4003) who were treated with infliximab and/or other medical therapies for IBD. Information will be collected on patient demographics, disease characteristics, clinical status, quality of life, medications, and dose and frequency of administration of infliximab, other biologics, and immune modulators.
Sampling Method: Non-Probability Sample
Enrollment: 4970 (Actual)
Dates: Start 2007-05-31 (Actual); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Obtain long-term safety and clinical status information on pediatric patients with IBD (ie, CD, UC, or indeterminate colitis [IC]). | This is a 20-year registry that has visits every 6 months.
  The objective of this registry is to obtain long-term safety and clinical status information on pediatric patients with IBD (ie, CD, UC, or IC).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Services, L.L.C. Clinical Trial, Study Director — Janssen Services, L.L.C.
Locations (62):
- United States (58):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Oakland, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Portland, Maine
  - Boston, Massachusetts
  - Newton, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Boys Town, Nebraska
  - Las Vegas, Nevada
  - Manchester, New Hampshire
  - Mays Landing, New Jersey
  - Morristown, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Lake Success, New York
  - Mineola, New York
  - New York, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Williamsville, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (4):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Toronto, Ontario